CLINICAL TRIAL: NCT02544906
Title: Propofol Versus Dexmedetomidine for Prevention of Sevoflurane Agitation in Recipients of Living Donor Liver Transplantation
Acronym: Agitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AlRefaey Kandeel (Other)
Responsible Party: Sponsor-Investigator, AlRefaey Kandeel, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LTx 7
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Liver Transplantation
Keywords: recipients
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): No drugs will be given. the emergence agitation will be monitored and recorded
- Propofol group (Experimental): Propofol at dose of 1 mg/kg over 5 minutes will be started before extubation. the emergence agitation will be monitored and recorded
  Interventions: Drug: Propofol
- dexmedetomedine group (Experimental): dexmedetomedine at dose of .5 mic/kg over 5 minutes will be started before extubation. the emergence agitation will be monitored and recorded
  Interventions: Drug: dexmedetomedine

INTERVENTIONS:
Drug: Propofol — Infusion of propofol to prevent emergence agitation in liver transplanta recipients
  Arms: Propofol group
Drug: dexmedetomedine — Infusion of dexmedetomedine to prevent emergence agitation in liver transplanta recipients
  Arms: dexmedetomedine group

SUMMARY:
The use of propofol or dexmedetomedine for prevention of sevofurane emergence agitation in LDLT recipients

ELIGIBILITY:
Inclusion Criteria:

* All recipients of living donor liver transplantation

Exclusion Criteria:

* patient refusal Allergy to either propofol or dexmedetomediene CNS disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
incidence of emergence agitation in liver trasnplant recipients | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt